CLINICAL TRIAL: NCT05960981
Title: Effects of Parent-Mediated Intervention on Restricted and Repetitive Behaviors in Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sabri Hergüner (Other)
Responsible Party: Sponsor-Investigator, Sabri Hergüner, associate professor, Herguner Therapy Private Clinic
Organization: Herguner Therapy Private Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HergunerTheraPC
Record Dates: First submitted 2023-07-08; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder;; Social communication; Restricted and repetitive behavior; Parent mediated intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Communication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention grup (Experimental): The work is one-armed. It consists of only those in the intervention group. After the study was announced, informed consent was obtained from those who agreed to participate in the study. Afterwards, the participants filled out the Demographic Data Form, Repetitive Behavior Scale-Revised (RBS-R), Social Communication Checklist-Revised (SCC-R), Child Behavior Checklist-Dysregulation Profile (CBCL-DP) forms before the intervention program started. When the 8-week online group-based parent mediated intervention program was over, they filled out formsRepetitive Behavior Scale-Revised (RBS-R), Social Communication Checklist-Revised (SCC-R), Child Behavior Checklist-Dysregulation Profile (CBCL-DP) again in the first week.
  Interventions: Behavioral: Online-delivered Group-based Parent Mediated Intervention for Young Children with ASD

INTERVENTIONS:
Behavioral: Online-delivered Group-based Parent Mediated Intervention for Young Children with ASD — The program consists of eight weekly 2-hour group sessions, with each group consisting of 8 to 10 families. During the sessions, supervisors present the strategies to the parents and explain how to integrate them into their interactions with their children. Sample videos are shown to illustrate the strategies, and group discussions allow parents to discuss their application. In the second half of each session, the parents' recorded videos are watched, and supervisors provide feedback on whether the strategies were accurately implemented. At the end of each session, supervisors address any questions the parents may have.

SUMMARY:
Our primary aim in the study is to investigate the effect of an online group-based 8-week parent-mediated intervention program targeting social communication on restrictive repetitive behaviors. Our second aim is to investigate the factors affecting the change in restrictive repetitive behavior. Our hypotheses are that after completing the 8-week online group-based parent-mediated intervention program, the participants' social interaction skills will increase, their restrictive repetitive behaviors will decrease, and their emotion regulation problems will decrease.

DETAILED DESCRIPTION:
Repetitive motor movements, preoccupations with objects, strict adherence to routines and rituals, and a resistance to change are all examples of restricted repetitive behaviors (RRBs). These behaviors are not exclusive to autism spectrum disorder (ASD) and can also be observed in children with intellectual disabilities and typically developing children. However, children with ASD tend to exhibit RRBs more frequently, severely, and intensely.

Studies have shown that as typically developing children improve their language and social interaction skills, the frequency of RRBs tends to decrease. On the other hand, research involving children with ASD has demonstrated that RRBs are associated with a decline in social interaction abilities. However, there are also studies suggesting that RRBs are unrelated to social communication skills. Anxiety has been found to be connected to RRBs in children with ASD, and one study even identified emotion regulation problems as the strongest predictor of RRBs.

RRBs can consume a significant amount of time, limit opportunities for social interactions, and hinder the acquisition of new skills in children. They can also have a negative impact on family functioning and well-being. Parents often find managing RRBs to be the most stressful and challenging aspect of dealing with ASD. Unfortunately, research on restricted repetitive behaviors is limited, with a primary focus on pharmacological treatments and behavioral interventions that predominantly utilize single-case designs. Various strategies have been employed with some success to address RRBs, such as blocking, interrupting, and redirecting for lower-order RRBs, as well as cognitive behavioral therapy and differential reinforcement strategies for higher-order RRBs. However, managing RRBs remains a significant challenge for parents, as the available interventions have limited effectiveness.

RRBs create considerable difficulties for both children with ASD and their families. In this study, we aim to investigate the impact of an 8-week online group-based parent-mediated intervention on restricted repetitive behaviors. Additionally, we will explore the factors that influence the improvement of these behaviors. This research endeavor is expected to provide valuable insights and contribute to the existing knowledge on effectively managing RRBs. The findings have the potential to benefit both professionals and parents by equipping them with enhanced coping strategies. Furthermore, this study will contribute to the expansion of scientific literature regarding the effects of parent-mediated interventions on addressing RRBs, thereby advancing our understanding in this area.

ELIGIBILITY:
Inclusion Criteria:

* the child had a confirmed clinical diagnosis of ASD,
* the child was aged between 2 and 6 years,
* the parents were able to speak and read Turkish sufficiently,
* parents agreed not to start any other new intensive interventions during the study,
* same parent could attend each session

Exclusion Criteria:

* a medical condition that impacted development (e.g., Fragile X, Down syndrome, tuberous sclerosis
* enrolment in any other parent-mediated intervention(s) during the study

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Change in restricted repetitive behavior | baseline and 2.5 months
  We examined the effect of intervention on RRBs by using the change in Repetitive Behavior Scale-Revised (RBS-R) scores. After the intervention program, whether there were significant changes in the total scores and subscales of Repetitive Behavior Scale-Revised (RBS-R) was determined by the paired t test if it met the normal distribution conditions, and the Wilcoxon test if it did not meet the normal distribution conditions.Repetitive Behavior Scale-Revised (RBS-R): The RBS-R is a 43-item parent rating scale. All items are rated on a four-point Likert scale of severity; the higher the scores, the more severe the conditions (i.e., 0 = behavior does not occur, 1 = behavior occurs and is a mild problem, 2 = behavior occurs and is a moderate problem, 3 = behavior occurs and is a severe problem). The scale can be scored between 0-129.
Chance in social communication | baseline and 2.5 months
  We examined the effect of intervention on social cominication by using the change in Social Communication Checklist-Revised (SCC-R) scores. After the intervention program, whether there were significant changes in the total scores and subscales of Social Communication Checklist-Revised (SCC-R) was determined by the paired t test if it met the normal distribution conditions, and the Wilcoxon test if it did not meet the normal distribution conditions.Social Communication Checklist-Revised (SCC-R): The SCC-R is a 70-item checklist.They are summed for domain scores and a Total Score. Respondents indicate whether a child uses each skill, "Rarely/Not Yet (1)," "Sometimes, but not consistently (2)," or "Usually, at least 75% of the time (3)". The total score would then be between 70 and 215. An increase in the Total Score means that social communication skills have increased.
change in emotion disregulation | baseline and 2.5 months
  We examined the effect of intervention on emotion disregulation by using the change in Child Behavior Checklist-Dysregulation Profile(CBCL-DP) scores. After the intervention program, whether there were significant changes in the total scores and subscales of Child Behavior Checklist-Dysregulation Profile (CBCL-DP) was determined by the paired t test if it met the normal distribution conditions, and the Wilcoxon test if it did not meet the normal distribution conditions.Child Behavior Checklist-Dysregulation Profile (CBCL-DP): CBCL 1.5-5 is a 99-item. The CBCL-DP score is computed by the sum of the Attention, Aggression, and Anxious/Depressed subscales of the CBCL 1.5-5. The item is marked as 0 if the child does not have it, 1 if it is sometimes or somewhat true for the child, and 2 if it is very true or often true. An increase in total score means that emotional dysregulation is exacerbated.

SECONDARY OUTCOMES:
Factors predicting change in restrictive repetitive behaviors | baseline and 2.5 months
  The difference between the total units of the scale at the baseline assessment and the total units of the scale 2.5 months later was calculated arithmetically.To partition the variance associated with change observed in RRBs (measured by Repetitive Behavior Scale-Revised )over the intervention, we performed step-wise hierarchical regression analysis by including change observed in social communication (measured by Social Communication Checklist-Revised), emotion regulation (measured by Child Behavior Checklist-Dysregulation Profile), and age as independent variables.

CONTACTS AND LOCATIONS:
Overall Officials: Sabri Hergüner, assoc.Prof., Study Director — Hergüner Therapy Private Clinic
Locations (1):
- Hergüner Therapy Private Clinic, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD in one publication that forms the basis of the results
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data can be shared 6 months after the study is published
Access Criteria: Assoc.Prof. Dr. Sabri Hergüner will review the requests.